CLINICAL TRIAL: NCT00004196
Title: A Multicenter Trial of Adjuvant Interferon Alfa-2b for Melanoma Patients With Early Lymph Node Metastasis Detected by Lymphatic Mapping and Sentinel Lymph Node Biopsy
Brief Title: Interferon Alfa-2b in Treating Patients With Melanoma and Early Lymph Node Metastasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CDR0000067439; UAB-9735; UAB-F970925009; NCI-G99-1654; RPCI-DS-99-14
Record Dates: First submitted 2000-01-21; First posted 2003-01-27 (Estimated); Last update posted 2014-01-20 (Estimated); Status verified 2013-04

CONDITIONS: Melanoma (Skin)
Keywords: stage I melanoma; stage II melanoma; stage III melanoma
MeSH Terms: conditions — Melanoma | interventions — Interferon-alpha; Observation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- AI (Experimental): Patients with metastasis in a single sentinel node with no evidence of extracapsular extension and no metastatic disease in nonsentinel nodes are randomized to 1 of 2 treatment arms. Patients receive adjuvant high-dose interferon alfa-2b IV 5 days a week for 4 weeks, then subcutaneously 3 times a week for 48 weeks
  Interventions: Biological: recombinant interferon alfa
- Arm AII (Experimental): Patients with metastasis in a single sentinel node with no evidence of extracapsular extension and no metastatic disease in nonsentinel nodes are randomized to 1 of 2 treatment arms. Observational arm: Patients with metastases in more than one sentinel node with evidence of extracapsular extension or metastasis in any nonsentinel node receive adjuvant high-dose interferon alfa-2b as in arm AI.
  Interventions: Biological: recombinant interferon alfa; Drug: Observation
- Arm BI (Experimental): Patients with positive sentinel node(s) by PCR analysis are randomized to one of three treatment arms. Patients undergo observation. Patients are followed every 3 months for 2 years, every 4 months for 1 year, every 6 months for 2 years, and then annually thereafter.
  Interventions: Drug: Observation
- Arm B II (Experimental): Patients with positive sentinel node(s) by PCR analysis are randomized to one of three treatment arms. Patients undergo lymph node dissection. Patients are followed every 3 months for 2 years, every 4 months for 1 year, every 6 months for 2 years, and then annually thereafter.
  Interventions: Procedure: lymphangiography
- Arm BIII (Experimental): Patients with positive sentinel node(s) by PCR analysis are randomized to one of three treatment arms. Patients undergo lymph node dissection followed by adjuvant high-dose interferon alfa-2b IV 5 days a week for 4 weeks.
  Patients are followed every 3 months for 2 years, every 4 months for 1 year, every 6 months for 2 years, and then annually thereafter.
  Interventions: Biological: recombinant interferon alfa; Procedure: lymphangiography

INTERVENTIONS:
Biological: recombinant interferon alfa
  Arms: AI; Arm AII; Arm BIII
Procedure: lymphangiography
  Arms: Arm B II; Arm BIII
Drug: Observation
  Arms: Arm AII; Arm BI

SUMMARY:
RATIONALE: Interferon alfa-2b may interfere with the growth of cancer cells.

PURPOSE: Randomized phase III trial to study the effectiveness of interferon alfa-2b in treating patients who have melanoma with early lymph node metastasis.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of regional lymphadenectomy with or without adjuvant high-dose interferon alfa-2b on disease-free survival and overall survival of patients with invasive cutaneous melanoma with early or submicroscopic sentinel lymph node metastasis detected by histology or immunohistochemistry or by polymerase chain reaction (PCR).
* Compare the effect of lymphadenectomy vs observation on disease-free survival and overall survival of patients with submicroscopic sentinel lymph node metastasis detected only by PCR.
* Determine the recurrence rate and survival of patients with submicroscopic sentinel lymph node metastasis detected only by PCR.
* Determine the positive and negative predictive value of reverse transcriptase PCR analysis of sentinel lymph nodes and peripheral blood to identify patients at risk for recurrence and death.

OUTLINE: This is a randomized, multicenter study. Patients in the randomized portions of Protocols A and B are stratified according to tumor thickness (1-2 mm vs 3-4 mm vs greater than 4 mm) and tumor ulceration (yes vs no).

All patients undergo wide local tumor excision with lymphatic mapping and sentinel node biopsy. Patients with tumors with ambiguous drainage patterns undergo lymphoscintigraphy prior to tumor excision. Patients with evidence of metastatic melanoma in the sentinel node(s) by routine histology, serial sectioning, or immunohistochemistry and who have undergone a prior regional lymph node dissection proceed to protocol A.

* Protocol A: Patients with metastasis in a single sentinel node with no evidence of extracapsular extension and no metastatic disease in nonsentinel nodes are randomized to 1 of 2 treatment arms.

  * Arm I: Patients receive adjuvant high-dose interferon alfa-2b IV 5 days a week for 4 weeks, then subcutaneously 3 times a week for 48 weeks.
  * Arm II: Patients undergo observation. Patients with metastases in more than one sentinel node with evidence of extracapsular extension or metastasis in any nonsentinel node receive adjuvant high-dose interferon alfa-2b as in arm I.

Patients with no evidence of sentinel node(s) metastases by routine histology, serial sectioning, and immunohistochemistry and are negative by polymerase chain reaction (PCR) analysis are observed.

* Protocol B: Patients with positive sentinel node(s) by PCR analysis are randomized to one of three treatment arms.

  * Arm I: Patients undergo observation.
  * Arm II: Patients undergo lymph node dissection.
  * Arm III: Patients undergo lymph node dissection followed by adjuvant high-dose interferon alfa-2b IV 5 days a week for 4 weeks.

Patients are followed every 3 months for 2 years, every 4 months for 1 year, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 3,000 patients will be accrued for this study within 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed invasive cutaneous melanoma

  * Breslow thickness at least 1.0 mm
  * Primary site must be on head, neck, trunk or extremity
  * No more than 90 days since biopsy
* Protocol A:

  * One or more sentinel lymph nodes with histologic or immunohistochemical evidence of metastatic melanoma
  * Prior regional lymph node dissection
* Protocol B:

  * Sentinel lymph nodes with no histologic or immunohistochemical evidence of metastatic melanoma
  * Sentinel lymph node positive by reverse transcriptase polymerase chain reaction
* No prior wide local excision of the primary tumor with a margin greater than 1.5 cm
* No primary melanoma involving the eye or mucous membranes
* No clinical evidence of satellite lesions or intransit, regional nodal, or distant metastases
* No second primary invasive melanoma
* No prior surgery in the region of the primary draining nodal basin that would disrupt normal lymphatic drainage patterns (e.g., skin grafts, tissue transfers or flaps, or lymph node dissections)

PATIENT CHARACTERISTICS:

Age:

* 18 to 70

Performance status:

* Karnofsky 70-100%

Life expectancy:

* At least 10 years

Hematopoietic:

* WBC at least 3,000/mm^3
* Absolute granulocyte count at least 1,500/mm^3
* Platelet count at least 70,000/mm^3
* Hemoglobin at least 10.0 g/dL

Hepatic:

* Bilirubin less than 2.0 mg/dL
* SGOT/SGPT less than 3 times upper limit of normal (ULN)
* Alkaline phosphatase less than 3 times ULN
* No severe decompensated liver disease (e.g., cirrhosis or autoimmune hepatitis)
* No other significant liver disease that would preclude study participation

Renal:

* Creatinine normal

Cardiovascular:

* No cardiovascular disease (e.g., angina or congestive heart failure)
* No myocardial infarction within the past year
* No tachyarrhythmias

Pulmonary:

* No severe debilitating pulmonary disease (e.g., chronic obstructive pulmonary disease)

Other:

* No hypersensitivity to interferon alfa-2b or related compounds or any component of the injection
* No major depression or other major psychiatric illness
* No thyroid disorder with thyroid function that is not maintained within the normal range with medications
* No autoimmune disease
* No primary or secondary immunodeficiencies
* No severe diabetes mellitus prone to ketoacidosis
* No significant retinal abnormalities
* No evidence of infection
* No other malignancy within the past 5 years except basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or stage I laryngeal cancer
* No other medical condition that would preclude study participation
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after the study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior immunotherapy

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* At least 6 months since prior oral or parenteral steroids

Radiotherapy:

* No prior radiotherapy

Surgery:

* See Disease Characteristics
* No prior organ transplantation

Other:

* At least 6 months since prior immunosuppressants
* No concurrent immunosuppressants resulting from prior organ transplantation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 1999-10; Primary Completion 2004-10 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marshall M. Urist, MD, Study Chair — University of Alabama at Birmingham
Locations (4):
- United States (4):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York